CLINICAL TRIAL: NCT06915896
Title: Predictive Variables of Outcome in Subjects With Chronic Rachialgia Referred to Different Pathways of Physiotherapy: Multicenter Prospective Study
Brief Title: Predictive Variables of Outcome in Subjects With Chronic Rachialgia Referred to Different Pathways of Physiotherapy.
Acronym: PRE-CBP
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Francesca Cecchi, Professor, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: PRE-CBP
Record Dates: First submitted 2025-03-13; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Chronic Non-Specific Low Back Pain; Chronic Non-specific Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic spinal pain patients attending public health rehabilitation pathways

SUMMARY:
The aim of this study is to investigate the predictive value of various biopsychosocial variables on the outcomes of subjects with chronic spinal pain undergoing public health rehabilitation pathways. Secondly, the study aims to assess the reliability of certain questionnaires, classified as Patient-Reported Outcome Measures (PROMs), which are frequently used in the evaluation of spinal pain but whose metric properties have not yet been established. These objectives will be pursued through two comprehensive assessment sessions (before and after rehabilitation), a re-test session immediately before rehabilitation (to evaluate the reliability of the questionnaires in stable subjects), and two follow-up assessments at 3 and 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age of majority;
* Medical diagnosis of nonspecific low back pain or nonspecific neck pain;
* Chronic symptoms, present for at least 6 months;
* Waiting for rehabilitation in a public health pathways
* Signature of informed consent to participate in the study and processing of personal data.

Exclusion Criteria:

* Subjects with cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with nonspecific spinal pain waiting for rehabilitation in public health pathways.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | Second sessions (T1), after 3 month from enrollment
  The Neck Disability Index (NDI) is a questionnaire that helps assess how neck pain affects a person's daily life. It consists of 10 sections, each exploring a specific aspect, such as the intensity of pain, the ability to dress and bathe, lift weights, read, concentrate, work, drive, sleep, and engage in leisure activities.
  For each section, the patient must choose one answer from six options, with a score ranging from 0 to 5. The lowest score indicates no difficulty, while the highest indicates pain so severe that it makes it impossible to perform the activity.
  In the end, by adding up the scores from all sections, a maximum score of 50 points is obtained. The higher the score, the greater the disability related to neck pain.
  (only on neck pain patients)
Roland and Morris Disability Questionnaire | Third session (T2), after 6 months from enrollment
  The Roland Morris Disability Questionnaire is used to assess low back pain. It consists of 24 questions directed at the patient regarding their ability or limitation in performing the 24 activities listed, which are typically difficult for a patient with low back pain to carry out. Additionally, the phrase "Due to the back..." has been added to the questions to distinguish limitations caused by lower back pain from those caused by other factors. The administration time is about 5 minutes.
  For each activity, the patient must give a score of 0 if the activity is not limited, or 1 if they have difficulty due to back pain. The total score ranges from 0 to 24.
  (only on low back pain patients)
Neck Disability Index | Third session (T2), after 6 months from enrollment
  The Neck Disability Index (NDI) is a questionnaire that helps assess how neck pain affects a person's daily life. It consists of 10 sections, each exploring a specific aspect, such as the intensity of pain, the ability to dress and bathe, lift weights, read, concentrate, work, drive, sleep, and engage in leisure activities.
  For each section, the patient must choose one answer from six options, with a score ranging from 0 to 5. The lowest score indicates no difficulty, while the highest indicates pain so severe that it makes it impossible to perform the activity.
  In the end, by adding up the scores from all sections, a maximum score of 50 points is obtained. The higher the score, the greater the disability related to neck pain.
  (only on neck pain patients)
Roland and Morris Disability Questionnaire | Second sessions (T1), after 3 month from enrollment
  The Roland Morris Disability Questionnaire is used to assess low back pain. It consists of 24 questions directed at the patient regarding their ability or limitation in performing the 24 activities listed, which are typically difficult for a patient with low back pain to carry out. Additionally, the phrase "Due to the back..." has been added to the questions to distinguish limitations caused by lower back pain from those caused by other factors. The administration time is about 5 minutes.
  For each activity, the patient must give a score of 0 if the activity is not limited, or 1 if they have difficulty due to back pain. The total score ranges from 0 to 24.
  (only on low back pain patients)
Neck Disability Index | T0, at the enrollment
  The Neck Disability Index (NDI) is a questionnaire that helps assess how neck pain affects a person's daily life. It consists of 10 sections, each exploring a specific aspect, such as the intensity of pain, the ability to dress and bathe, lift weights, read, concentrate, work, drive, sleep, and engage in leisure activities.
  For each section, the patient must choose one answer from six options, with a score ranging from 0 to 5. The lowest score indicates no difficulty, while the highest indicates pain so severe that it makes it impossible to perform the activity.
  In the end, by adding up the scores from all sections, a maximum score of 50 points is obtained. The higher the score, the greater the disability related to neck pain.
  (only on neck pain patients)
Roland and Morris Disability Questionnaire | T0, at the enrollment
  The Roland Morris Disability Questionnaire is used to assess low back pain. It consists of 24 questions directed at the patient regarding their ability or limitation in performing the 24 activities listed, which are typically difficult for a patient with low back pain to carry out. Additionally, the phrase "Due to the back..." has been added to the questions to distinguish limitations caused by lower back pain from those caused by other factors. The administration time is about 5 minutes.
  For each activity, the patient must give a score of 0 if the activity is not limited, or 1 if they have difficulty due to back pain. The total score ranges from 0 to 24.
  (only on low back pain patients)
TAMPA SCALE of KINESIOPHOBIA | re-test at baseline
  test-retest relative reliability (intraclass correlation coefficient) of TAMPA SCALE of KINESIOPHOBIA (only on neck pain patients).
  It's a self-report questionnaire designed to assess pain beliefs and pain-related fear of movement in subjects with musculoskeletal disorders
PAIN AWARENESS AND VIGILANCE QUESTIONNAIRE | re-test at baseline
  test-retest relative reliability (intraclass correlation coefficient) of PAIN AWARENESS AND VIGILANCE QUESTIONNAIRE (only on neck pain patients).
  It is a self-report questionnaire to measure attention to pain
PITTSBURGH SLEEP QUALITY INDEX | re-test at baseline
  test-retest relative reliability (intraclass correlation coefficient) of PITTSBURGH SLEEP QUALITY INDEX (only on neck pain patients). It is a rating scale developed for the purpose of providing a reliable, valid and standardized measure of sleep quality.
TAMPA SCALE of KINESIOPHOBIA | re-test at baseline
  test-retest absolute reliability (minimal detectable change (mdc) 95) of TAMPA SCALE of KINESIOPHOBIA (only on neck pain patients).
  It's a self-report questionnaire designed to assess pain beliefs and pain-related fear of movement in subjects with musculoskeletal disorders.
PAIN AWARENESS AND VIGILANCE QUESTIONNAIRE | re-test at baseline
  test-retest absolute reliability (minimal detectable change (mdc) 95) of PAIN AWARENESS AND VIGILANCE QUESTIONNAIRE (only on neck pain patients).
  It is a self-report questionnaire to measure attention to pain
PITTSBURGH SLEEP QUALITY INDEX | re-test at baseline
  test-retest absolute reliability (minimal detectable change (mdc) 95) of PITTSBURGH SLEEP QUALITY INDEX (only on neck pain patients). It is a rating scale developed for the purpose of providing a reliable, valid and standardized measure of sleep quality.

SECONDARY OUTCOMES:
Pain Intensity | T0, at the enrollment
  Numeric Pain Raiting scale 0-10
Pain Intensity | Second sessions (T1), after 3 month from enrollment
  Numeric Pain Raiting scale 0-10
Pain Intensity | Third session (T2), after 6 months from enrollment
  Numeric Pain Raiting scale 0-10
Health Related Quality of Life | T0, at the enrollment
  Short-Form 12 (SF12)
Self-reported change | Third session (T2), after 6 months from enrollment
  Global rating of Change Scale
Self-reported change | Second sessions (T1), after 3 month from enrollment
  Global rating of Change Scale
Self-reported change | T0, at the enrollment
  Global rating of Change Scale
Medication Use | Third session (T2), after 6 months from enrollment
  yes/no
Medication Use | Second sessions (T1), after 3 month from enrollment
  yes/no
Medication Use | T0, at the enrollment
  yes/no
Pain Frequency | Third session (T2), after 6 months from enrollment
  0-7 in a week
Pain Frequency | Second sessions (T1), after 3 month from enrollment
  0-7 in a week
Pain Frequency | T0, at the enrollment
  0-7 in a week
Health Related Quality of Life | Third session (T2), after 6 months from enrollment
  Short-Form 12 (SF12)
Health Related Quality of Life | Second sessions (T1), after 3 month from enrollment
  Short-Form 12 (SF12)
Pain Catastrophizing Scale (PCS) | T0, at the enrollment
  The Pain Catastrophizing Scale (PCS) is a measurement scale based on a 13-item self-completion questionnaire designed to assess catastrophizing pain-related thoughts in adults with or without chronic pain.
  (only for patients with cervicalgia)
Pain Catastrophizing Scale (PCS) | Second sessions (T1), after 3 month from enrollment
  The Pain Catastrophizing Scale (PCS) is a measurement scale based on a 13-item self-completion questionnaire designed to assess catastrophizing pain-related thoughts in adults with or without chronic pain.
  (only for patients with cervicalgia)
Pain Catastrophizing Scale (PCS) | Third session (T2), after 6 months from enrollment
  The Pain Catastrophizing Scale (PCS) is a measurement scale based on a 13-item self-completion questionnaire designed to assess catastrophizing pain-related thoughts in adults with or without chronic pain.
  (only for patients with cervicalgia)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No